CLINICAL TRIAL: NCT04228757
Title: A Clinical Study Assessing Efficacy of an Herbal Blend on Menopausal Symptoms and Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: i-Health, Inc. (Industry)
Collaborators: ObvioHealth (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OBVIO-DSM-003
Record Dates: First submitted 2019-12-20; First posted 2020-01-14 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Menopause
Keywords: Nutritional Supplement

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled intervention
Who Masked: Participant, Care Provider, Investigator
Masking Description: A unique ID number will be assigned by ClaimIt to each enrolled subject and associated with the correct study product kit number; this number will be used throughout the study. Both the study product and placebo will be labeled identically except for kit number and will be distinguishable only by the individual participant ID and kit number.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Herbal Blend (Experimental): A phytoestrogen herbal blend
  Interventions: Dietary Supplement: phytoestrogen herbal blend
- Placebo (Placebo Comparator): Tablet without active ingredients
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: phytoestrogen herbal blend — phytoestrogen herbal blend
  Arms: Investigational Herbal Blend
Other: Placebo — Tablet without active ingredients
  Arms: Placebo

SUMMARY:
This 12-week study is a randomized, placebo-controlled study assessing the efficacy of an herbal blend on menopausal symptoms and quality of life.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate changes in menopause symptoms after taking an herbal supplement daily for 12 weeks compared to placebo (a tablet that does not have active ingredients). This is a remote study, meaning all study data will be collected via the ClaimIt app, with the exception of a screening lab appointment and a Week 12 lab appointment.Participants will be asked to report on study compliance and respond to a series of questionnaires relating to symptoms of menopause, hot flashes, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Females between 40 and 65 years of age
* Report experiencing moderate to severe menopausal symptoms, characterized as including all of the following:

  * Total Score of 11 or greater on the Greene Climacteric Scale (GCS) Questionnaire
  * Self-reported frequent hot flashes experienced (estimated minimum of 28 during the past week, or an average of a minimum of 4 in a typical day)
  * Absence of a regular menstrual cycle, defined as either: an irregular cycle for at least 6 months, or the absence of menses for 3 or more months
* Agreement to maintain current level of physical activity throughout the study period
* Willingness and ability to follow the procedures of the study
* Willingness and ability to provide informed consent

Exclusion Criteria:

* Participant with a Body Mass Index (BMI) ≥ 30mg/kg2
* Participant who has had both ovaries removed
* Women who are pregnant, breastfeeding, or planning on becoming pregnant during the course of the study
* A history of breast cancer or a positive mammogram
* A history of uterine cancer or an abnormal pap smear
* Abnormal vaginal bleeding (not related to menstrual irregularity)
* Liver disease
* A history of clinically diagnosed depression that a medical professional recommended should be medically treated
* A history of clinically diagnosed hypertension (systolic of 140 mmHg or greater or diastolic of 90 mmHg or greater)
* Hyperthyroidism determined by thyroid stimulating hormone (TSH) screening
* Any unstable medical condition as determined by the Principal Investigator (PI)
* Any significant clinical or laboratory abnormality identified by the PI
* Any change in the use of dietary supplements in the 2-month prior to enrollment
* The use of any product indicated for menopause symptoms in the 2 months prior to enrollment including: prescription drugs (e.g. estrogen/progestins), over-the-counter supplements (e.g. black cohosh, soy isoflavones, evening primrose oil, phytoestrogens, etc), or a significant change in diet to include more soy foods.
* The use of any psychiatric drugs in the 6 months prior to enrolling
* Self-reported abuse of drugs or alcohol
* Any smoking of cigarettes, vaping or e-cigarettes, or consumption of other tobacco products within the past 6 months
* Planned donation of blood during or up to 30 days after completion of the study
* An allergy to any ingredient in the herbal blend product or placebo
* A sensitivity to botanical extracts
* Previous participation in a clinical research study less than 30 days prior to randomization to a treatment group
* Any other condition that in the investigator's opinion may adversely affect the participant's ability to complete the study, or may pose a significant risk to the participant

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 130 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2020-04-04 (Estimated); Study Completion 2020-04-04 (Estimated)

PRIMARY OUTCOMES:
Overall Menopausal Symptoms | 12 weeks
  Change from baseline in global menopausal symptoms assessed by the Greene Climacteric Questionnaire at Week 12.
  The Greene Climacteric Questionnaire is a 21-item validated questionnaire that provides a measurement of global menopause symptoms, grouping questions into psychological, physical, vasomotor, and sexual domains. Participants answer on a 4-point scale. Each response is given a numerical value from 0 to 3 points respectively, and the sum total of their 21-point responses is calculated as their GCS score.

SECONDARY OUTCOMES:
Overall Menopausal Symptoms | 8 weeks
  Change from baseline in global menopausal symptoms assessed by Greene Climacteric questionnaire at weeks 2, 4 and 8.
  The Greene Climacteric Questionnaire is a 21-item validated questionnaire that provides a measurement of global menopause symptoms, grouping questions into psychological, physical, vasomotor, and sexual domains. Participants answer on a 4-point scale. Each response is given a numerical value from 0 to 3 points respectively, and the sum total of their 21-point responses is calculated as their GCS score.
Incidence/severity of hot flash episodes | 12 weeks
  Change from baseline in frequency of hot flash episodes as measured by self-report of incidence of hot flashes at week 2, 4, 8, and 12, considering:
  * Total number of episodes
  * Number of episodes per category of intensity: mild, moderate, severe and very severe
Feelings of fatigue | 12 weeks
  Change from baseline in feelings of fatigue as measured by Chalder Fatigue Scale questionnaire scores at weeks 4, 8, and 12.
  The CFS is an 11-point questionnaire that provides a numerical value for overall symptoms of fatigue. Participants are asked to answer about their experience of fatigue related symptoms on a 4-point scale including "Less than usual", "No more than usual", "More than usual" and "Much more than usual" on the first 10 questions. On the final question the options are "Better than usual", "No worse than usual", "Worse than usual" and "Much worse than usual". Each score is given a numerical score of 0-3 respectively, and a total calculated as the sum of the 11 responses.
Health-related quality of life (EQ-VAS) | 12 weeks
  Change from baseline in health-related quality of life as measured by the EuroQol visual analogue scale (EQ-VAS) at weeks 2, 4, 8, and 12.
  The EQ-VAS is a questionnaire that requires participants to report self-perception of how good their health is that day on a 100-point visual analogue scale.
Vaginal dryness | 12 weeks
  Change from baseline in self-reported vaginal dryness on a five-point scale as measured by response to a study-specific questionnaire item at weeks 2, 4, 8, and 12
Perception of wellness | 12 weeks
  Participant perception of wellness after 12 weeks of supplementation, as documented by listed responses to open-ended questions in a study-specific questionnaire.

OTHER OUTCOMES:
Blood biomarkers | 12 weeks
  Chemistry Panel including liver enzymes and CBC
Incidence of AEs | 12 weeks
  Incidence of Adverse Events (AEs) observed during the treatment period, classified by the investigator as to intensity, relationship to study product/protocol, and seriousness

CONTACTS AND LOCATIONS:
Overall Officials: Parth Shah, MD, Principal Investigator — ObvioHealth
Locations (1):
- ObvioHealth, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Utian WH, Archer DF, Bachmann GA, Gallagher C, Grodstein Fn, Heiman JR, Henderson VW, Hodis HN, Karas RH, Lobo RA, Manson JE, Reid RL, Schmidt PJ, Stuenkel CA; North American Menopause Society. Estrogen and progestogen use in postmenopausal women: July 2008 position statement of The North American Menopause Society. Menopause. 2008 Jul-Aug;15(4 Pt 1):584-602. doi: 10.1097/gme.0b013e31817b076a. PMID 18580541
- [Background] Chlebowski RT, Kuller LH, Prentice RL, Stefanick ML, Manson JE, Gass M, Aragaki AK, Ockene JK, Lane DS, Sarto GE, Rajkovic A, Schenken R, Hendrix SL, Ravdin PM, Rohan TE, Yasmeen S, Anderson G; WHI Investigators. Breast cancer after use of estrogen plus progestin in postmenopausal women. N Engl J Med. 2009 Feb 5;360(6):573-87. doi: 10.1056/NEJMoa0807684. PMID 19196674
- [Background] Rossouw JE, Anderson GL, Prentice RL, LaCroix AZ, Kooperberg C, Stefanick ML, Jackson RD, Beresford SA, Howard BV, Johnson KC, Kotchen JM, Ockene J; Writing Group for the Women's Health Initiative Investigators. Risks and benefits of estrogen plus progestin in healthy postmenopausal women: principal results From the Women's Health Initiative randomized controlled trial. JAMA. 2002 Jul 17;288(3):321-33. doi: 10.1001/jama.288.3.321. PMID 12117397
- [Background] Lethaby A, Marjoribanks J, Kronenberg F, Roberts H, Eden J, Brown J. Phytoestrogens for menopausal vasomotor symptoms. Cochrane Database Syst Rev. 2013 Dec 10;2013(12):CD001395. doi: 10.1002/14651858.CD001395.pub4. PMID 24323914